CLINICAL TRIAL: NCT06139146
Title: The Effectiveness of Muscle Energy Technique Combined With Strengthening of Deep Neck Flexors With and Without Core Stability Exercise in Upper Cross Syndrome Patients. A Randomized Control Trial
Brief Title: The Effectiveness of Muscle Energy Technique Combined With Strengthening of Deep Neck Flexors With and Without Core Stability Exercise in Upper Cross Syndrome Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, DR. SUNDUS NAZ, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2695
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Upper Cross Syndrome; Forward Head Posture
Keywords: core stability; muscle energy technique; core stability exercise; Goniometer; craniovertebral (CV) angle
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Control (Experimental): A moist heat pack for 15-20 minutes MET of the upper trapezius, levator scapula and pectoral Major muscles Strengthening exercise of deep neck flexors
  Interventions: Other: Muscle energy technique (MET)
- Group B Experimental (Experimental): A moist heat pack for 15-20 minutes Core stability exercises MET of the upper trapezius, levator scapula and pectoral Major muscles Strengthening exercise of deep neck flexors
  Interventions: Other: Core stability exercises:

INTERVENTIONS:
Other: Muscle energy technique (MET) — MET treatment protocol of pectoral major:
  The patient's position was supine lying. Starting with the position which took the affected fibres to just short of their restriction barrier, the patient introduced a light contraction involving adduction of the arm against resistance from the therapist for 7-10 seconds. As the patient exhaled the therapist stretched across the new barrier.
  MET treatment protocol of upper trapezius:
  The patient moved the stabilized shoulder in a shrug motion toward the ear, and the ear toward the shoulder, with a light resistance (20% of possible strength). The contraction was sustained for 7-1 0 seconds MET treatment protocol of levator scapula The patient was in a supine position, with the hand supinated and the arm of the side to be tested extended alongside the trunk.
  Strengthening of deep neck flexors: Patient was instructed to his nod head to flatten the neck's curve. 10 reps for 10 sec.
  Other Names: Strengthening of deep neck flexors; Moist heat pack
  Arms: Group A Control
Other: Core stability exercises: — Warm up: The cat and camel stretches
  Exercises:
  * It included Crook lying, abdominal bracing, and 10 second - 20 repetitions (reps).
  * Crook lying, abdominal Bracing with leg lifts holding the position for 3 second for 10 reps.
  * Crook lying, abdominal Bracing with bridging with 10 reps with a 10 second hold.
  * It included a Quadruped position with abdominal bracing for 10 s - 10 reps
  * Quadruped position arm lifts with abdominal bracing 10 reps on each side.
  * Quadruped position leg lifts with abdominal bracing 10 reps on each side.
  * Quadruped position alternate arm and leg lifts with abdominal bracing holding position for 3 s - 10 reps on each side.
  * The curl-up in hook lying, Fold arms across the torso. Lift shoulder blades off the ground. 1 to 2 seconds holds - 10 reps.
  * Side plank on knees; holding position for 10 s - 5 reps .
  Arms: Group B Experimental

SUMMARY:
Upper cross syndrome (UCS) is a common muscles related postural disorder which is increasing every new day that is affecting the health related quality of life. It is most prevalent amongst the individuals who work at computers or laptops, or on desks.

The UCS is caused by poor posture. Weak core musculature leads to poor body posture causing chronic degenerative changes and disturbing body alignment and body equilibrium. Core stability exercises (CSE) are a good strategy to improve body posture. The purpose of this study is to determine the effects of muscle energy technique (MET) combined with the strengthening of deep neck flexors with and without core stability exercise to manage Upper Cross Syndrome (UCS) patients.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted at the Dow University of Health Sciences Ojha campus in Karachi, Pakistan. Those patients who fulfill the criteria will be enrolled in physiotherapy OPD and general OPD. Then they will be randomized into two groups as per the random allocation sheet for treatment. Pre- and post-intervention assessment for pain, functional disability, and range of motions will be done by visual analog scale (VAS), neck disability index (NDI), and goniometer.

Analysis of pre- and post-intervention measure analysis will be performed using SPSS version 21.The Sampling technique will be Nonprobability purposive sampling with Sample size of 70 participants (35 in each group).

Intervention: The Participant will be divided into two groups as per the random allocation sheet for treatment. In Group A, the control group will receive a moist heat pack for 20 minutes then muscle energy technique (MET) of the upper trapezius, levator scapula, and pectoralis muscles (major and minor) and strengthening exercise of deep neck flexors. In Group B, the experimental group will receive the same treatment session as the control group along with the Core stability exercise. There will be 12 sessions for each patient, 6 sessions regularly in the 1st week and then 3 sessions per week for the next 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were diagnosed or referred with UCS
* The participant with the age of 18 - 45 years old.
* Both male and female.
* Craniovertebral angle less than 48.
* Restricted cervical range of motion.

Exclusion Criteria:

* • Participants who were diagnosed with: Inflammatory/Rheumatoid Arthritis , neurological disorders, History of trauma or fracture with cervical spine, Cervical spine surgery or trauma or any spinal Congenital deformities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (change is being assessed) | Baseline and 3 weeks.
  The primary outcome is self-reported neck pain on visual analog scale. VAS validate subjective measure for acute and chronic pain. The VAS consists of a line that is 10 cm long, with two end points that stand for 0 (meaning "no pain") and 10 (meaning "pain as bad as it could be"). VAS is the most reliable among numerical rating scale (NRS) and verbal rating scale (VRS)

SECONDARY OUTCOMES:
Craniovertebral angle (change is being assessed) | Baseline and 3 weeks.
  The craniovertebral angle measure by Goniometric method which is accepted as reliable method. Measurement will be perform in standing position. The intersection of a horizontal line that goes through the C7 spinous process and a line that connects the middle of the tragus of the ear to the skin overlying the C7 spinous process is known as the craniovertebral angle. With inter-rater reliability for the measurements has been found to be good (Cronbach's Alpha = 0.893).
Neck Disability Index (change is being assessed) | Baseline and 3 weeks.
  Neck disability index (NDI) will use to assess how neck pain affected daily living activities. The urdu version of NDI is an easy-to-understand and free to use, intra-class correlation coefficient (ICC2,1) revealed excellent test-retest reliability for all items with a Cronbach's alpha of 0.90, and good content validity.
Cervical range of motions (change is being assessed) | Baseline and 3 weeks.
  It measure by using Goniometer and goniometric measurements had established validity and reliability. Previous studies found that the intra-tester reliability was greater than the inter-tester reliability in both clinical and research setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. SUNDUS NAZ, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No